CLINICAL TRIAL: NCT04579471
Title: Prevalence and Outcome of SARS-CoV-2 Infection in Solid Organ and Hematopoietic Cell Transplant Recipients: The COVITRA Study
Brief Title: Prevalence and Outcome of SARS-CoV-2 Infection & COVID-19 in Transplant Recipients: The COVITRA Study
Acronym: COVITRA
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other); Hasselt University (Other); Ziekenhuis Oost-Limburg (Other); Jessa Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: s64036
Record Dates: First submitted 2020-10-06; First posted 2020-10-08 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Covid19; SARS-CoV Infection; Transplantation Infection
Keywords: covid19; SARS-CoV Infection; transplantation
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Collection and storage plasma samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Transplanted patients: All patients who underwent solid organ or hematopoietic cell transplantation at UZ Leuven
  Interventions: Diagnostic Test: SARS-CoV-2 IgG
- Transplanted patients with past SARS-CoV-2 infection: Transplanted patients with past SARS-CoV-2 infection will be followed for one year (at month 3, 6 and 12 after the initial study visit) to assess durability of IgG positivity
  Interventions: Diagnostic Test: SARS-CoV-2 IgG
- Transplanted patients without past SARS-CoV-2 infection: 100 transplanted patients without past SARS-CoV-2 infection will be followed for one year (at month 3, 6 and 12 after the initial study visit) to assess durability of IgG positivity and as control for the transplanted patients with WITH past SARS-CoV-2 infection
  Interventions: Diagnostic Test: SARS-CoV-2 IgG

INTERVENTIONS:
Diagnostic Test: SARS-CoV-2 IgG — Collection of clinical variables, assessment of IgG antibodies for SARS-CoV-2, plasma collection for translational immunology studies

SUMMARY:
This project will provide novel data using a large cohort of more than 3000 transplanted patients. Risk and protective factors for SARS-CoV-2 infection and COVID-19 disease severity will be identified. The proportion of patients who develop antibodies after infection will be revealed. In this way the presence of these antibodies can be evaluated as a test for prior infection. Our study additionally will demonstrate how long these antibodies remain present and whether they are protective against a new infection.

ELIGIBILITY:
Inclusion Criteria:

* all patients who underwent solid organ or hematopoietic cell transplantation at UZ Leuven and who give informed consent

Exclusion Criteria:

* age under 18 years

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients who underwent solid organ or hematopoietic transplantation at UZ Leuven and who give informed consent
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence and risk-factors for SARS-CoV-2 infection | inclusion during 4 months
  Prevalence and risk-factors for SARS-CoV-2 infection
Prevalence and risk-factors for COVID-19 | inclusion during 4 months
  Prevalence and risk-factors for COVID-19

SECONDARY OUTCOMES:
Durability of IgG positivity | 12 months
  Durability of IgG positivity/immunity

CONTACTS AND LOCATIONS:
Overall Officials: Jef Verbeek, MD, PhD, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Undecided